CLINICAL TRIAL: NCT04291547
Title: Computerised Behavioural Activation Programme for the Treatment of Depression in Young People: Feasibility Study
Brief Title: Computerised Behavioural Activation for Young People With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of York (Other)
Responsible Party: Principal Investigator, Lucy Tindall, Principal Investigator, University of York
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 270172
Record Dates: First submitted 2020-02-25; First posted 2020-03-02 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Low Mood; Depression
Keywords: Young people
MeSH Terms: conditions — Consciousness Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computerised Behavioural Activation Programme (Experimental): All recruited young people will be given the BALM (Behavioural Activation for Low Mood) programme to work through
  Interventions: Device: BALM

INTERVENTIONS:
Device: BALM — An online Behavioural Activation programme for young people with mild to moderate low mood/depression. The programme comprises 10 treatment sessions lasting 30 to 45 minutes

SUMMARY:
The primary aim of this non-randomised feasibility study is to 1) examine the acceptability of a newly developed computerised Behavioural Activation programme (BALM) in treating young people experiencing low mood/depression and 2) assess the feasibility of undertaking a pilot Randomised Controlled Trial (RCT) of the intervention.

DETAILED DESCRIPTION:
Approximately 20% of adolescents will have had at least one depressive episode by the age of 18 making depression one of the leading causes of illness and disability in young people. Although receiving effective treatment is important, as few as 35% of young people seek help, with treatment-related issues (e.g. stigma, negative attitudes about help-seeking, accessibility, reluctance to engage one-to-one with a therapist, etc) outlined as reasons for this. Computerised therapies, which have increased availability and accessibility, reduced stigma and can be delivered in a format attractive to many young people may avoid some of these barriers and provide a more effective treatment option for young people.

Behavioural Activation (BA) - a type of talking therapy focused on increasing liked activities has demonstrated effectiveness in treating depression in adults and, owing to this, is an evidence-based treatment for depression within NICE (2009) guidelines. Despite this, less research has examined its use with young people.

We have developed BALM (Behavioural Activation for Low Mood), an online BA programme designed for use with young people experiencing mild to moderate low mood or depression. The development of BALM was based upon the findings of a systematic review and a series of qualitative interviews and focus groups with young people and healthcare professionals.

Eligible young people will be referred to the programme via healthcare professionals working in local Child and Adolescent Mental Health Services and mental health practitioners based in local secondary schools.

The findings of this research will allow us to refine the intervention and the research methods we employ in preparation for a pilot randomised controlled trial (RCT) of the new treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 11 to 16 years at the date of consent
* Experiencing low mood or depression symptoms as defined by a score of ≥20 on the Mood and Feelings Questionnaire
* In agreement that their primary care provider and a parent/guardian can be informed of any concerns the lead researcher has about their wellbeing during participation

Exclusion Criteria:

* Within the normal range on the measure of depressive symptoms (i.e. attaining a score of ≤19 on the Mood and Feelings Questionnaire)
* Experiencing severe low mood or depression symptoms
* Having a comorbid mental health diagnosis of Bipolar Disorder or Psychosis.
* Non-English speaking (due to the small scope of this study, the option of providing translated versions of BALM and the outcome measures was not feasible)
* Deemed to be actively at risk of self harm or suicide
* Have no access to the internet and therefore no programme access

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of undertaking a pilot Randomised Controlled Trial of BALM by examining questionnaire response rates | 4 months
  Assessed by examining questionnaire response rates
Feasibility of undertaking a pilot Randomised Controlled Trial of BALM by examining the percentage of those eligible who consented | 4 months
  Assessed by examining the percentage of those eligible who consented to the study
Feasibility of undertaking a pilot Randomised Controlled Trial of BALM by examining number and reasons for withdrawal | 4 months
  Assessed by examining number and reasons for withdrawal
Feasibility of undertaking a pilot Randomised Controlled Trial of BALM by examining session attendance | 4 months
  Assessed by examining session attendance
To examine the acceptability of BALM in treating young people experiencing low mood/depression by examining session adherence | 4 months
  Assessed by examining session adherence
To examine the acceptability of BALM in treating young people experiencing low mood/depression by examining responses on an evaluation questionnaire | 4 months
  Assessed by examining responses on an evaluation questionnaire comprising 15 short questions

CONTACTS AND LOCATIONS:
Overall Officials: Barry Wright, Study Chair — University of York; Dean McMillan, Study Chair — University of York; Antonina Mikocka-Walus, Study Chair — Deakin University
Locations (1):
- Tees Esk and Wear Valleys NHS Foundation Trust, York, United Kingdom

IPD SHARING:
Plan to Share IPD: No